CLINICAL TRIAL: NCT01472705
Title: Long-Term Comparison of Everolimus-Eluting and Biolimus-Eluting Stents in All-Comer Patients
Brief Title: Everolimus- Versus Biolimus-Eluting Stents in All-Comers
Acronym: EverBio
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Stéphane Cook, Prof, Principal Investigator, University of Freiburg
Other Study IDs: 003-REP-CER-FR
Record Dates: First submitted 2011-08-30; First posted 2011-11-16 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting coronary stent; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- everolimus-eluting stents (EES): Second-generation everolimus-eluting stents (EES) have been shown to be superior to the first-generation paclitaxel eluting stents (PES) in terms of safety and efficacy.
- biolimus-eluting stents (BES): Third generation biolimus-eluting stents (BES) have been shown to be superior to the PES and non inferior to first-generation sirolimus eluting stents in terms of safety and efficacy.

SUMMARY:
This study sought to investigate safety and efficacy of biolimus-eluting stents (BES) with biodegradable polymer as compared with everolimus-eluting stents (EES) with durable polymer through 3 years of follow-up.

DETAILED DESCRIPTION:
A group of 814 consecutive patients undergoing percutaneous coronary intervention (PCI) was enrolled between 2007 and 2010, of which 527 were treated with EES and 287 with BES implantation. Clinical outcome was compared in 200 pairs using propensity score matching. The primary endpoint was a composite of death, myocardial infarction (MI) and target vessel revascularisation (TVR) at two-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* all patients with at least one BES or EES for de novo stenosis

Exclusion Criteria:

* patients with at least one non-study stent
* patients with both study stent
* patients with life expectancy < 3 years

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated at our institution with at least one BES or EES
Sampling Method: Probability Sample
Enrollment: 814 (Actual)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Composite of Death, Myocardial Infarction and Target Vessel Revascularization | up to 24 months
  The primary outcome is the above mentioned composite of adverse events in order to measure their cumulative incidence (i.e. the rate of occurrence of such events in the study population over a predefined time periode).

SECONDARY OUTCOMES:
Cardiovascular death | up to 24 months
Any Revascularization | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane P Cook, MD, Study Chair — University Fribourg; Mario Togni, MD, Study Director — University Fribourg; Markus Oberhänsli, MD, Principal Investigator — University Fribourg
Locations (1):
- Cardiology, university Fribourg Medical Center, Fribourg, Canton of Fribourg, Switzerland

REFERENCES:
- [Result] Puricel S, Oberhansli M, Guntern P, Lehmann S, Goy JJ, Arroyo D, Villeneuve H, Baeriswyl G, Stauffer JC, Togni M, Cook S. Long-term comparison of everolimus-eluting and biolimus-eluting stents. EuroIntervention. 2013 Jul;9(3):336-44. doi: 10.4244/EIJV9I3A55. PMID 23482296
- [Result] Arroyo D, Togni M, Puricel S, Gerard B, Sonja L, Corpataux N, Villeneuve H, Boute E, Stauffer JC, Goy JJ, Cook S. Comparison of everolimus-eluting and biolimus-eluting coronary stents with everolimus-eluting bioresorbable scaffold: study protocol of the randomized controlled EVERBIO II trial. Trials. 2014 Jan 7;15:9. doi: 10.1186/1745-6215-15-9. PMID 24398143